CLINICAL TRIAL: NCT03258307
Title: Comparison of Perilipin, Leptin, Adipolipin, Adiponectin, Resistin, Visfatin, Estrone Levels Derivated From Adipose Tissue Pre-postoperatively in Patient Diagnosed With Gynecological Malignancy Performed Omentectomy or Not
Brief Title: Comparison of Perilipin, Leptin, Adipolipin, Adiponectin, Resistin, Visfatin, Estrone Levels Pre-post Omentectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Isa Aykut Ozdemir, Head of Department of Gynecologic Oncology Bakirkoy Dr Sadi Konuk Training and Research Hospital, Istanbul Training and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 900
Record Dates: First submitted 2017-08-15; First posted 2017-08-23 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Gynecologic Cancer

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- omentectomy (Active Comparator): Preoperative
  Interventions: Other: Preoperative level
- Omentectomy (Other): Postoperative
  Interventions: Other: Preoperative level
- No omentectomy (Other): Preoperative post operative
  Interventions: Other: Preoperative level

INTERVENTIONS:
Other: Preoperative level — Blood sample
  Other Names: Postoperative level

SUMMARY:
Omentum is adipose tissue lying under inner anterior wall Omentectomy is routine procedure in treatment of gynecological malignancy especially ovarian cancer and some advanced stage endometrial cancer. Perilipin, Leptin, Adipolipin, Adiponectin, Resistin, Visfatin, Estrone secrete from adipose tissue. These regulate matabolic process.

We aimed comparison of Perilipin, Leptin, Adipolipin, Adiponectin, Resistin, Visfatin, Estrone levels derivated from adipose tissue pre-postoperatively in patient diagnosed with gynecological malignancy performed omentectomy or not

DETAILED DESCRIPTION:
Omentum is adipose tissue lying under inner anterior wall Omentectomy is routine procedure in treatment of gynecological malignancy especially ovarian cancer and some advanced stage endometrial cancer. Perilipin, Leptin, Adipolipin, Adiponectin, Resistin, Visfatin, Estrone secrete from adipose tissue. These regulate matabolic process.

We aimed comparison of Perilipin, Leptin, Adipolipin, Adiponectin, Resistin, Visfatin, Estrone levels derivated from adipose tissue pre-postoperatively in patient diagnosed with gynecological malignancy performed omentectomy or not. Blood sample will study after 4000 rpm centrifugal for 10 minutes

ELIGIBILITY:
Inclusion Criteria:

* gynecologic malignancy, staging surgery with or without omentectomy

Exclusion Criteria:

* not accept inclusion to trial

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
with omentectomy group | 1 year
  Pre-postoperative levels of Perilipin, Leptin, Adipolipin, Adiponectin, Resistin, Visfatin, Estrone
No omentectomy group | 1 year
  Pre-postoperative levels of Perilipin, Leptin, Adipolipin, Adiponectin, Resistin, Visfatin, Estrone

CONTACTS AND LOCATIONS:
Locations (1):
- Bakirkoy Dr Sadi Konuk Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD will not share other researchers due to participant individual preference but when the research result publish researchers may obtain

REFERENCES:
- [Derived] Comba C, Ozdemir IA, Demirayak G, Erdogan SV, Demir O, Ozlem Yildiz G, Bulut H, Karakas S, Gulseren V, Afsar S, Gungorduk K. The effect of omentectomy on the blood levels of adipokines in obese patients with endometrial cancer. Obes Res Clin Pract. 2022 May-Jun;16(3):242-248. doi: 10.1016/j.orcp.2022.06.002. Epub 2022 Jun 11. PMID 35701296